CLINICAL TRIAL: NCT05728099
Title: Effect of SpiroGym Mobile Application in Expiratory Muscle Strength Training in Patients With Parkinson's Disease: a Double Blind Randomised Control Trial
Brief Title: Effect of SpiroGym App in Patients With Parkinson's Disease
Acronym: RespPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Martin Srp, Ph.D., Chief physiotherapist of the rehabilitation section in General University Hospital Prague, General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 223/20 S-IV
Record Dates: First submitted 2023-01-20; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Expiratory muscle strength training; Adherence
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the experimental or the active control group. A simple computer-generated random allocation sequence was completed before study initiation.
Who Masked: Participant, Outcomes Assessor
Masking Description: During the whole study protocol, patients did not receive information about testing the SpiroGym app. They will receive information that we are testing two types of expiratory muscle strength training programs. Outcomes assessors are blinded to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expiratory muscle strength training + SpiroGym application (Experimental): The experimental arm will undergo 24 weeks of expiratory muscle strength training coupled with SpiroGym app.
  Interventions: Device: Expiratory muscle strength training + SpiroGym application
- Expiratory muscle strength training (Active Comparator): The experimental arm will undergo 24 weeks of expiratory muscle strength training.
  Interventions: Device: Expiratory muscle strength training

INTERVENTIONS:
Device: Expiratory muscle strength training + SpiroGym application — Participants will performe an intensive home-based expiratory muscle training programme using an Expiratory Muscle Trainer (EMST150; Aspire Products, LLC, United States), which provide a pressure- threshold range from 30 to 150 cmH20. EMST therapy sessions will be completed at home on 5 days of the patients choosing per week. Participants will be instructed to perform five sets of five forceful expirations coupled with SpiroGym app. per training session for 8 weeks (intensive training period). For another 16 weeks (maintenance period) participants will be instructed to perform, at least twice per week, five sets of five forceful expirations coupled with SpiroGym app. per training session .
  Arms: Expiratory muscle strength training + SpiroGym application
Device: Expiratory muscle strength training — Participants will performe an intensive home-based expiratory muscle training programme using an Expiratory Muscle Trainer (EMST150; Aspire Products, LLC, United States), which provide a pressure- threshold range from 30 to 150 cmH20. EMST therapy sessions will be completed at home on 5 days of the patients choosing per week. Participants will be instructed to perform five sets of five forceful expirations per training session for 8 weeks (intensive training period). For another 16 weeks (maintenance period) participants will be instructed to perform, at least twice per week, five sets of five forceful expirations per training session. Participants will be given the practice log to track training adherence.
  Arms: Expiratory muscle strength training

SUMMARY:
Airway protective disorders, including swallowing (dysphagia) and cough (dystussia) are common in patients with Parkinson's disease (PD). Disturbances in these protective mechanisms increase the risk of aspiration pneumonia. In fact, aspiration pneumonia is the leading cause of death in individuals with PD. Expiratory muscle strength training (EMST) studies have reported significant improvements in the field of airway protective therapies. EMST represents a treatment that can be quantified and translated into functional outcomes that can directly improve functions related to coughing, swallowing, and speech in patients with PD. However, information about detraining outcomes presented in Troche et al. 2014 highlights the need for the development of long-term maintenance programs to sustain training gains following intensive periods of EMST, especially considering the progressive nature of PD. Low long-term adherence to home exercise is an important issue in many patient groups and may compromise treatment outcomes. In patients with PD, this is further compounded by a wide variety of neuropsychiatric symptoms, such as apathy and depression. Therefore, we developed a mobile phone-based visual feedback application (SpiroGym app.) to keep patients motivated to continue EMST following intensive periods of training. The usability of a SpiroGym app was tested in individuals with PD and the findings indicate that EMST coupled with SpiroGym app is feasible and potentially useful in PD patients. Present study aims to verify and extend the encouraging results of this study which showed a potential self-efficacy benefit of the SpiroGym application.

DETAILED DESCRIPTION:
Goal 1: To explore effect of the SpiroGym apllication on treatment adherence in 24weeks home expiratory strength training.

Hypothesis: Treatment adherence will be higher in the experimental group than in the active control group.

Goal 2: To explore self-efficacy effect of the SpiroGym aplication in expiratory muscle training.

Hypothesis: The SpiroGym application will increase self-eficacy for expiratory muscle strength training.

Goal 3: To explore additional visual feedback effect of the SpiroGym application to increase training effort compared with regular training without immediate visual feedback.

Hypothesis: Visual feedback of the SpiroGym application will increase training effort in expiratory muscle strength trainning which will be reflected in the MEP values at 8weeks assessment and 24weeks assessment.

Study design: a double blind randomised-controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinsons disease
* Stable dopaminergic medication (stable dose for at least 1 month)
* Patient in the risk of non-adherence to the home exercise program (SEHEPS questionnaire below 59 points)

Exclusion Criteria:

* Other neurological disorders
* Difficulty complying due to neuropsychological dysfunction (dementia with a score of less than 19 on the Montreal Cognitive Assessment)
* Breathing disorders or diseases
* Smoking in the past 5 years
* Uncontrolled hypertension

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Treatment adherence | Adherence for home exercise programs from baseline to end of the study (24 weeks)
  Adherence will be calculated by comparing the total amount of expiratory maneuvers recorded in the patient training logs (active control group) or in the SpiroGym application (experimental group) to the prescribed amount: 1000 manoeuvres during baseline to week 8 and 800 manoeuvres during weeks 8-24.

SECONDARY OUTCOMES:
Maximum expiratory pressure (MEP) | 1 week before baseline, baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks and 24 weeks
  MEP assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines. Assessments will be performed using a flanged rubber mouthpiece connected to a pressure manometer (Micro RPM, Micro Medical).The maximum value of three expiratory maneuvers that vary by less than 10%. However, results of published studies confirms a learning effect in the MEP measurements. In order to eliminate the learning effect, the patients will be examined twice within one week. The value from the second measurement will be taken as the baseline MEP value. Aditionaly to decrease the test's variability, a 'warm up session' will be incorporated prior to MEP measurements.
The Self-Efficacy scale for home exercise programs | baseline, 8 weeks
  The Self-Efficacy scale for home exercise programs is a tool for evaluating a patient's self-efficacy for home-based exercise programs. The minimum value is 0 and the maximum value is 72. Higher score mean higher self-efficacy for performing home exercise programs.

OTHER OUTCOMES:
MDS-Unified Parkinson's Disease Rating Scale: part III. | Baseline, 8 weeks and 24 weeks
  This portion of the scale assesses the motor signs of Parkinson´s disease. The minimum value is 0 and the maximum value is 132. Higher score mean The minimum value is 0 and the maximum value is 72. Higher score mean higher patient motor disability.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Srp, Ph.D., Principal Investigator — General University Hospital, Prague
Locations (1):
- General University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srp M, Korteova R, Kliment R, Jech R, Ruzicka E, Hoskovcova M. Expiratory Muscle Strength Training in Patients with Parkinson's Disease: A Pilot Study of Mobile Monitoring Application. Mov Disord Clin Pract. 2021 Aug 4;8(7):1148-1149. doi: 10.1002/mdc3.13313. eCollection 2021 Oct. No abstract available. PMID 34631956
- [Background] Reyes A, Castillo A, Castillo J. Effects of Expiratory Muscle Training and Air Stacking on Peak Cough Flow in Individuals with Parkinson's Disease. Lung. 2020 Feb;198(1):207-211. doi: 10.1007/s00408-019-00291-8. Epub 2019 Nov 12. PMID 31720808
- [Background] Troche MS, Curtis JA, Sevitz JS, Dakin AE, Perry SE, Borders JC, Grande AA, Mou Y, Vanegas-Arroyave N, Hegland KW. Rehabilitating Cough Dysfunction in Parkinson's Disease: A Randomized Controlled Trial. Mov Disord. 2023 Feb;38(2):201-211. doi: 10.1002/mds.29268. Epub 2022 Nov 7. PMID 36345090
- [Background] Troche MS, Rosenbek JC, Okun MS, Sapienza CM. Detraining outcomes with expiratory muscle strength training in Parkinson disease. J Rehabil Res Dev. 2014;51(2):305-10. doi: 10.1682/JRRD.2013.05.0101. PMID 24933728
- [Background] Palazzo C, Klinger E, Dorner V, Kadri A, Thierry O, Boumenir Y, Martin W, Poiraudeau S, Ville I. Barriers to home-based exercise program adherence with chronic low back pain: Patient expectations regarding new technologies. Ann Phys Rehabil Med. 2016 Apr;59(2):107-13. doi: 10.1016/j.rehab.2016.01.009. Epub 2016 Apr 1. PMID 27050664
- [Background] Chagraoui A, Boukhzar L, Thibaut F, Anouar Y, Maltete D. The pathophysiological mechanisms of motivational deficits in Parkinson's disease. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Feb 2;81:138-152. doi: 10.1016/j.pnpbp.2017.10.022. Epub 2017 Oct 31. PMID 29097256
- [Background] Picha KJ, Lester M, Heebner NR, Abt JP, Usher EL, Capilouto G, Uhl TL. The Self-Efficacy for Home Exercise Programs Scale: Development and Psychometric Properties. J Orthop Sports Phys Ther. 2019 Sep;49(9):647-655. doi: 10.2519/jospt.2019.8779. Epub 2019 Jul 10. PMID 31291552
- [Background] Claus I, Muhle P, Czechowski J, Ahring S, Labeit B, Suntrup-Krueger S, Wiendl H, Dziewas R, Warnecke T. Expiratory Muscle Strength Training for Therapy of Pharyngeal Dysphagia in Parkinson's Disease. Mov Disord. 2021 Aug;36(8):1815-1824. doi: 10.1002/mds.28552. Epub 2021 Mar 2. PMID 33650729
- [Background] Reyes A, Castillo A, Castillo J, Cornejo I, Cruickshank T. The Effects of Respiratory Muscle Training on Phonatory Measures in Individuals with Parkinson's Disease. J Voice. 2020 Nov;34(6):894-902. doi: 10.1016/j.jvoice.2019.05.001. Epub 2019 May 31. PMID 31155431
- [Background] Pitts T, Bolser D, Rosenbek J, Troche M, Okun MS, Sapienza C. Impact of expiratory muscle strength training on voluntary cough and swallow function in Parkinson disease. Chest. 2009 May;135(5):1301-1308. doi: 10.1378/chest.08-1389. Epub 2008 Nov 24. PMID 19029430
- [Background] Volianitis S, McConnell AK, Jones DA. Assessment of maximum inspiratory pressure. Prior submaximal respiratory muscle activity ('warm-up') enhances maximum inspiratory activity and attenuates the learning effect of repeated measurement. Respiration. 2001;68(1):22-7. doi: 10.1159/000050458. PMID 11223726